CLINICAL TRIAL: NCT04428086
Title: Open-Label, Fixed-Sequence Study in Solid Tumor Subjects to Investigate the Pharmacokinetic Interaction Between Apatinib and Transporter Substrates Rosuvastatin and Metformin.
Brief Title: A Pharmacokinetic Interaction Study Between Apatinib and Rosuvastatin or Metformin in Solid Tumor Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR-APTN-I-010
Record Dates: First submitted 2020-05-27; First posted 2020-06-11 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — apatinib; 26S proteasome non-ATPase regulatory subunit 13; Rosuvastatin Calcium; JPT1 protein, human; Metformin

STUDY DESIGN:
Intervention Model Description: Two arms Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assess PK effects of Apatinib on Rosuvastatin (Experimental): Participant will be administered a single oral dose of rosuvastatin 10 milligram (mg) on Day 1 and Day 7 and Apatinib at a dose of 250 mg once daily from Day 4 until Day 9.
  Interventions: Drug: Apatinib in arm1; Drug: Rosuvastatin
- Assess PK effects of Apatinib on Metformin (Experimental): Participant will be administered a single oral dose of metformin 500 milligram (mg) on Day 1 and Day 6 and Apatinib at a dose of 250 mg once daily from Day 3 until Day 7.
  Interventions: Drug: Apatinib in arm2; Drug: Metformin

INTERVENTIONS:
Drug: Apatinib in arm1 — Apatinib will be administered at a dose of 250 mg once daily from Day 4 to Day 9.
  Arms: Assess PK effects of Apatinib on Rosuvastatin
Drug: Rosuvastatin — Rosuvastatin will be administered as a single oral 10 milligram (mg) dose on Day 1 and Day 7.
  Arms: Assess PK effects of Apatinib on Rosuvastatin
Drug: Apatinib in arm2 — Apatinib will be administered at a dose of 250 mg once daily from Day 3 to Day 7.
  Arms: Assess PK effects of Apatinib on Metformin
Drug: Metformin — Metformin will be administered as a single oral 500 mg on Day 1 and Day 6.
  Arms: Assess PK effects of Apatinib on Metformin

SUMMARY:
The primary objective of the study was to assess investigate the pharmacokinetic effects of Apatinib on Rosuvastatin or Metformin.

The secondary objective of the study was to assess the safety of Apatinib alone or Rosuvastatin/Metformin alone or concomitant medication.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to enter the study:

1. Age: 18-70 years old (Include both values);
2. Patients with histopathologically or cytologically confirmed advanced solid tumor(except primary gastrointestinal tumors or metastatic gastrointestinal tumors and primary hepatocellular tumors) , not necessary to have measurable lesions;
3. The standard systemic treatment plan for tumors is ineffective, or intolerable, or there is no recurrence and metastasis after adjuvant chemotherapy and radiotherapy after surgery;
4. ECOG PS score: 0-1;
5. Expected survival ≥ 3 months;
6. Adverse reactions caused by the subject receiving other treatments have recovered (recovered to ≤ grade 1 according to NCI-CTCAE 5.0, except for hair loss), more than 4 weeks after receiving radiotherapy or surgery or receiving other cytotoxic drugs or cell growth inhibitor.
7. Major organs must function normally, meeting the following criteria:

   I. Haematology (no blood transfusion or blood products within the last 14 days, not corrected with G-CSF or other hematopoietic colony-stimulating factors):
   1. HB≥100 g/L;
   2. ANC≥1.5×109/L;
   3. PLT≥90×109/L;

   II. Blood biochemistry:
   1. TBIL≤ 1.25×ULN;
   2. ALT and AST≤2.5×ULN;
   3. ALP≤2.5×ULN;
   4. Serum Cr ≤ 1.5 × ULN or endogenous CrCl ≥ 60 mL/min (Cockcroft-Gault formula);
   5. Albumin > 30 g/L;

   III. Urine protein inspection:

   a. Urinary routines suggest that urine protein <++. If urinary protein ≥ ++, the quantification of urinary protein in 24 hours should be ≤1.5 g;
8. Agree to abstinence or take effective contraception during the study and for at least 8 weeks after the last study drug administration
9. Sign the ICF voluntarily, have good compliance, corporate with follow-up visits, and follow the study requirements.

Exclusion Criteria:

Subjects meeting any one of the followings will be excluded in this study:

1. Patients with gastrointestinal diseases that affect the use or absorption of drugs, such as gastric cancer or intestinal cancer, unable to swallow, chronic diarrhea, intestinal obstruction, large stomach or total gastrectomy, or within 6 months before the first medication Patients with abdominal fistula, gastrointestinal perforation or abdominal abscess;
2. Active (without medical control) brain metastases, cancerous meningitis, spinal cord compression patients, or imaging CT or MRI examination at screening to find diseases of the brain or pia mater
3. Presence of clinically symptomatic third space fluid (e.g. large pleural fluid or ascites) that cannot be controlled by drainage or other methods;
4. Patients with hypertension, or patients with a history of hypertension
5. Patients with NYHA Class III-IV cardiac insufficiency or left ventricular ejection fraction (LVEF) < 50% by echocardiography; uncontrolled arrhythmias (QTc interval ≥ 450 ms in males and ≥ 470 ms in females);
6. During the study period, patients should be used drugs that may lead to prolonged QTc interval (such as antiarrhythmic drugs, quinidine, disopyramide, procainamide, sotalol, amiodarone, etc.)
7. Patients with abnormal coagulation function (INR > 1.5 or prothrombin time (PT) > ULN + 4 s or APTT > 1.5 ULN)
8. Patients with clinically significant bleeding or clear bleeding tendency within 3 months prior to the first dose, such as coughing up blood, hemoptysis, GI bleeding, hemorrhagic gastric ulcer, or baseline fecal occult blood (FOB) ++ and above. Gastroscopy is required for patients with FOB (+) and no surgical resection of primary gastric tumor. In case of ulcerative gastric cancer, patients are not enrolled due to a risk of acute gastrointestinal hemorrhage;
9. Events of arterial/venous thrombosis within 6 months prior to the first dose, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, brain infarction), deep vein thrombosis, and pulmonary embolism;
10. Known hereditary or acquired hemorrhage and thrombophilia (such as hemophilia, coagulopathy, thrombocytopenia, hypersplenism, etc.);
11. Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or similar drugs;
12. Have undergone major surgery or with severe traumatic injury, fracture, or ulcer within 4 weeks prior to the first dose; There is no previous wound healing.
13. Use of study drugs in other clinical trials within 4 weeks prior to the first dose;
14. Drugs that is CYP3A inhibitor, or the transporter BCRP or MATE1 inhibitor, or drugs that affect gastric acid secretion, or Chinese herbal medicines within 2 weeks before the first dose; use the drug that is metabolic enzyme CYP3A inducer within 4 weeks before the first dose
15. Infectious disease screening (hepatitis B virus surface antigen, hepatitis C virus antibody, Treponema pallidum antibody and human immunodeficiency virus antibody) positive
16. History of immunodeficiency, with acquired, congenital immunodeficiency disease, or history of organ transplantation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-08-22 (Actual); Study Completion 2021-08-22 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Up to Day 10
  The Cmax is the maximum observed concentration
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) | Up to Day 10
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) | Up to Day 10
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | through study completion, an average of 35 or 37 days in two groups.
  An adverse event is any untoward medical occurrence in a patient or clinical study participant criteria

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: Undecided